CLINICAL TRIAL: NCT02124876
Title: Accommodating for Residual Limb Fluid Volume Change
Acronym: AM-PM
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Joan Sanders, Professor, University of Washington
Other Study IDs: STUDY00002557; R01HD060585 (NIH)
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Diurnal Residual Limb Fluid Volume Fluctuation
Keywords: amputee; prosthetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Transtibial amputees

SUMMARY:
The purpose of this study is to quantify residual limb fluid volume changes between morning and afternoon hours, and to determine if fluid volume change is correlated with activity.

ELIGIBILITY:
Inclusion Criteria:

* transtibial amputation
* at least 18 months after amputation surgery
* ability to walk on a treadmill and stand for 90 seconds

Exclusion Criteria:

* skin breakdown on the residual limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Transtibial amputee currently using prosthetic limbs
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06-06 (Actual); Study Completion 2014-06-06 (Actual)

PRIMARY OUTCOMES:
Residual limb fluid volume | 1 day

SECONDARY OUTCOMES:
Duration of walking and moving | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States